CLINICAL TRIAL: NCT00898898
Title: Analyses of c-Myc (MYC) and Topoisomerase II Alpha (TOP2A) Copy Number Aberrations; MYC, Insulin-like Growth Factor Receptor-1 (IGF-1R) and PTEN Protein Expressions; and Phosphatidylinositol 3' Kinase (PIK3) Gene Mutations in N9831 Primary Breast Tumors
Brief Title: Studying Tissue Samples From Women With Breast Cancer Who Were Treated on Clinical Trial NCCTG-N9831
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCCTG N9831-ICSC; NCCTG-N9831-ICSC; CDR0000593349 (Registry Identifier: PDQ (Physician Data Query)); NCI-2009-00687 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; HER2-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue (FFPE whole block sections and TMA sections)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Arm I: Tissue samples from protocol NCCTG-N9831 are obtained for immunohistochemistry and fluorescence in situ hybridization analysis of MYC, IGF- 1R, PTEN, and TOP2A genes. Exons 9 and 20 of PIK3CA gene are amplified via polymerase chain reaction; mutations in exons 9 and 20 of PIK3CA gene are identified.
  Interventions: Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Other: diagnostic laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is looking at tissue samples from women with breast cancer who were treated on clinical trial NCCTG-N9831. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the association between the primary breast tumor protein expression of MYC, IGF-1R, and PTEN and disease-free survival (DFS) in patients randomized on clinical trial NCCTG-N9831.

II. To determine the association between the primary breast tumor amplification status of MYC and TOP2A and DFS in patients randomized on NCCTG-N9831.

III. To determine the association between the primary breast tumor mutation status of PIK3 and DFS in patients randomized on NCCTG-N9831.

SECONDARY OBJECTIVES:

I. To determine the association between the primary breast tumor marker protein expression/amplification/mutation status of the aforementioned markers and overall survival in patients randomized on NCCTG-N9831.

II. To investigate the predictive potential of multiple marker analyses on DFS and overall survival using multivariate analysis.

III. To determine the correlation between the protein expression and amplification status of MYC in patients randomized on NCCTG-N9831.

IV. To determine the correlation between marker protein expression/amplification/mutation status and known clinicopathological characteristics of the tumors.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with breast cancer and treated on clinical trial NCCTG-N9831

  * Randomized to treatment
* HER-2 positive disease
* Whole tissue blocks and/or tissue microarray sections available
* Hormone receptor status:

  * ER/PR status known
* Any menopausal status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with primary HER2 positive breast cancer which received doxorubicin and cyclophosphamide (AC) followed by paclitaxel with or without trastuzumab.
Sampling Method: Non-Probability Sample
Enrollment: 2837 (Actual)
Dates: Start 2000-05 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Levels of primary breast tumor protein expression of MYC, IGF-1R, and PTEN assessed using standard immunohistochemical (IHC) procedures | Baseline
Levels of primary breast tumor amplification status of MYC and TOP2A assessed using standard fluorescence in situ hybridization (FISH) assays | Baseline
Levels of primary breast tumor mutation status of PIK3 assessed using molecular digestion followed by HPLC separation | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Derived] Perez EA, Jenkins RB, Dueck AC, Wiktor AE, Bedroske PP, Anderson SK, Ketterling RP, Sukov WR, Kanehira K, Chen B, Geiger XJ, Andorfer CA, McCullough AE, Davidson NE, Martino S, Sledge GW, Kaufman PA, Kutteh LA, Gralow JR, Harris LN, Ingle JN, Lingle WL, Reinholz MM. C-MYC alterations and association with patient outcome in early-stage HER2-positive breast cancer from the north central cancer treatment group N9831 adjuvant trastuzumab trial. J Clin Oncol. 2011 Feb 20;29(6):651-9. doi: 10.1200/JCO.2010.30.2125. Epub 2011 Jan 18. PMID 21245420